CLINICAL TRIAL: NCT01649713
Title: Tolerability and Immunogenicity Study of Fluval AB Suspension for Injection (Trivalent, Seasonal Influenza Vaccine, Active Ingredient Content: 15 ugHA/Strain/0.5mL) in Adult and Elderly Subjects
Brief Title: Yearly Licence Tolerability and Immunogenicity Study of Fluval AB Seasonal Influenza Vaccine to be Used in the 2012/2013 Vaccination Season
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Fluval AB-H-YL2012; 2012-002379-32 (EudraCT Number)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Influenza
Keywords: Fluval AB; influenza; vaccine; immunization; infections
MeSH Terms: conditions — Influenza, Human; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluval AB vaccination (Experimental): In this uncontrolled, open, multi-centre immunogenicity and tolerability study subjects will be enrolled into one vaccination group and will be vaccinated by a single injection of Fluval AB suspension for injection.
  Interventions: Drug: Fluval AB vaccination

INTERVENTIONS:
Drug: Fluval AB vaccination — Vaccination with Fluval AB suspension for injection

SUMMARY:
This is a yearly licence tolerability and immunogenicity study of Fluval AB suspension for injection (trivalent, seasonal influenza vaccine, active ingredient content: 15 μgHA/strain/0.5mL) in adult and elderly subjects to assess immunogenicity of a single intramuscular injection of Fluval AB suspension for injection, as measured by haemagglutination inhibition (HI) test, and to evaluate safety and tolerability (incidence of adverse events) of a single intramuscular injection of Fluval AB suspension for injection.

DETAILED DESCRIPTION:
For the 2011-2012 vaccination season the following influenza virus strains were recommended to be included in the influenza vaccines:

* A/California/7/2009(H1N1)-like virus,
* A/Perth/16/2009(H3N2)-like virus,
* B/Brisbane/60/2008-like virus.

For the 2012-2013 season the following strains were recommended (Amended EU Recommendations for the Seasonal Influenza Vaccine Composition for the Season 2012/2013, EMA/CHMP/BWP/140597/2012):

* A/California/7/2009(H1N1)-like virus,
* A/Victoria/361/2011(H3N2)-like virus,
* B/Wisconsin/1/2010-like virus.

Since the A/H3N2 and the B virus strains were changed, a yearly licence clinical study have to be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons aged 18 to 59 years, elderly persons aged ≥60 years from both sexes, mentally competent;
* Are in good health (as determined by vital signs and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known adequately treated clinically significant organ or systemic diseases (e.g. asthma or diabetes), such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study;
* Female volunteers aged 18-59 years (i.e. participants of childbearing potential) with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method or abstinence throughout the trial and not become pregnant for the duration of the study.
* Capability of participants to understand and comply with planned study procedures;
* Participants provide written informed consent prior to initiation of study procedures;
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy, breast feeding or positive urine pregnancy test at baseline prior to vaccination. Female subjects who are able to bear children but not willing to use an acceptable contraception method for the duration of the study.
* Known hypersensitivity to eggs, chicken protein, thiomersal, formaldehyde, gentamycin, ciprofloxacin, neomycin, vancomycin or any other component of the vaccine;
* History of Guillain-Barré syndrome;
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine;
* Serious disease, such as cancer, autoimmune disease, advanced arteriosclerotic disease, complicated diabetes mellitus, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure;
* Immunosuppressive therapy within 36 months prior to vaccination;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids;
* Receipt of immunostimulants;
* Receipt of parenteral immunoglobulin, blood products and/or plasma derivate within 3 months prior to vaccination;
* Suspected or known HIV, HBV or HCV infection;
* Acute disease and/or axillary temperature ≥37oC within 3 days prior to vaccination;
* Vaccine therapy within 4 weeks prior to vaccination;
* Influenza vaccination (any kind) within 6 months prior to vaccination;
* Experimental drug therapy within 4 weeks prior to vaccination;
* Concomitant participation in another clinical study;
* Any condition which, in the opinion of the investigator, may interfere with the evaluation of the study;
* Past or current psychiatric disease of the volunteer that upon judgement of the investigator may have effect on the objective decision-making of the volunteer;
* Alcohol or drug abuse of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Assessment of immunogenicity measures in comparison to criteria specified in CPMP/BWP/214/96 | 21-28 days after immunization
  To assess immunogenicity of a single intramuscular injection of Fluval AB suspension for injection (trivalent, seasonal influenza vaccine, active ingredient content: 15 μgHA/0.5mL of seasonal A/H1N1, A/H3N2 and B influenza antigens each), as measured by haemagglutination inhibition (HI) test in comparison to criteria specified in CPMP/BWP/214/96.

SECONDARY OUTCOMES:
To evaluate safety and tolerability (incidence of adverse events) of a single intramuscular injection of Fluval AB suspension for injection. | From Day 0 until 21-28 days after immunization
  Safety and tolerability will be assessed in comparison to available safety and tolerability data on Fluval AB suspension for injection:
  * number and percentage of subjects with at least one local reaction between Day 0 and Day 21-28.
  * number and percentage of subjects with at least one systemic reaction between Day 0 and Day 21-28.
  * number and percentage of subjects with at least one adverse reaction between Day 0 and Day 21-28.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitta Kozma, MD, Study Director — Omninvest Ltd.; Ferenc Tamás, MD, Principal Investigator — District Doctor's Office, Pilisvörösvar, Hungary
Locations (3):
- Hungary (3):
  - District Doctor's Office, Budapest
  - District Doctor's Office, Pilisvörösvar
  - District Doctor's Office, Szentendre